CLINICAL TRIAL: NCT05240716
Title: Assessing the Usefulness of Functional Electrical Stimulation Program on Tibial Nerve for Rehabilitation of Chronic Stroke Patients
Brief Title: Functional Electrical Stimulation on Tibial Nerve in Stroke Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Melisa Taborda, Principal Investigator, University of Gran Rosario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FES on TN in stroke
Record Dates: First submitted 2022-01-31; First posted 2022-02-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Chronic Stroke
Keywords: Functional electrical stimulation; Tibial Nerve stimulation; Chronic stroke; Hemiparetic gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES program (Experimental)
  Interventions: Other: FES program

INTERVENTIONS:
Other: FES program — 8 weeks intervention. 3 sessions per week. Previous to the intervention, volunteers will familiarize with the electrical stimulation by receiving three trials of the stimuli. Electrical current intensity will be set for each volunteers, with the capacity of generating a muscle contraction without inducing discomfort in the volunteer. During the FES program, patient in standing position will perform a step, while electrical current stimulation will be applied to the skin over the tibial nerve on the contralateral of the stimulation side. The FES will be delivered during the paretic plantarflexor activation according to the gait cycle. The FES session will consist of 5-minutes stimulation blocks with breaks between blocks (total session time: 30 minutes). For safety reasons, a physical therapist will supervise all the FES intervention sessions.

SUMMARY:
Hemiparetic gait is one of the most common consequences after stroke. This impairment has a detrimental effects on the patients lies, limiting their social participation. Previous studies have shown that there is a direct relationship between triceps surae activation and gait speed in stroke patients, that is, higher triceps surae muscle activation are correspond to greater gait speed. Then, it can be hypothesized that therapies focused in strengthening the triceps surae also improves the patient gait. It has been shown that Functional Electrical Stimulation (FES) can improve triceps surae activation when applied on healthy subjects. However, it has not been yet explored in chronic stroke patients. Therefore, the aim of this study is to assess whether a FES program over tibial nerve contributes to the rehabilitation of the gait in chronic hemiparetic stroke patients. This study present a prospective interventional design, based on non-probabilistic sampling for convenience, and comprising a total of 15 volunteers with ischemic stroke of both genders and aged between 18 and 70 years old. Volunteers will be recruited from hospitals and private rehabilitation centres, and must be currently engaged in a conventional rehabilitation program. The study will consist of twenty-four sessions, with a frequency of three sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging between 18 to 70 years.
* Subjects with chronic ischemic stroke (more than 12 months of evolution)
* Ability to walk 20 mts. without third-party assistance.
* Hemiparesis with weakness and spasticity in the triceps surae.

Exclusion Criteria:

* Previous injury on paretic lower limb
* Soft tissue or joint retraction limiting ankle range of motion (ROM)
* Severe peripheral nervous system compromise
* Electronic devices that could be altered by the use of FES (e.g. cardiac pacemaker)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in gait velocity | Baseline and week 8 (after 24 sessions of intervention)
  A 10 metres walk test will be performed to asses gait velocity.

SECONDARY OUTCOMES:
Change in maximal isometric strength | Baseline, immediately after first session and week 8 (after 24 sessions of intervention)
  To assess maximal isometric strength of dorsiflexor muscles, volunteers will performed 3 maximum repetitions of 6 seconds of isometric dorsiflexion. Force will be quantified using a load cell (maximum tension-compression = 200 Kgf, accuracy 0.1 Kgf, maximum measurement error = 0.33%; Equipo Biomédico Miotec ™, Porto Alegre, RS, Brazil), and this cell will be placed on a rigid surface and strapped to the volunteer's foot. In addition, the recorded force will be synchronised with the electromyograph to evaluate the isometric tensile strength. During this assessment, volunteers will be in supine position with the assessed lower limb extended on the stretcher.
Change in Spasticity | Baseline, immediately after first session and week 8 (after 24 sessions of intervention)
  The Modified Ashworth scale will be performed with volunteers in supine position, and the assessed lower limb extended on the stretcher. Passive stretching of the triceps surae will be applied at a constant speed from the position of maximum plantarflexion to the maximum possible dorsiflexion. Scores range from 0 to 4. A score of 0 indicates no resistance, and 4 indicates rigidity.
Change in muscle activity | Baseline, immediately after first session and week 8 (after 24 sessions of intervention)
  Surface electromyography (sEMG) will be recorded to assess activation of the tibialis anterior muscle. Four EMG channels will be acquired using commercial device (Miotec Suite ™, Biomedical Equipment, Porto Alegre, RS, Brazil). The electrodes (Ag/AgCl, with a centre-to-centre distance of 2 cm) will be align parallel to the muscle fibres of the tibialis anterior muscle, according to the recommendations of the International Society of Electrophysiology and Kinesiology (ISEK http://www.isek-online.org). A reference electrode will be placed on the lateral malleolus. Prior to electrode placement, the skin will be shaved and cleaned with cotton and 70% alcohol, in order to minimize skin impedance. The electromyographic recordings will be performed in the supine position, with the assessed leg extended and the opposite leg flexed at 70º with plantar support (measured by a goniometer).
Change in cortical electrical activity | Baseline and week 8 (after 24 sessions of intervention)
  Electroencephalography (EEG) will be recorded during active movement of the affected lower limb using a BIOAMP electroencephalography instrument (UNER, Oro Verde, Entre Ríos, Argentina), using a cap with 15 electrodes distributed according to the international 10-20 system. The volunteer will be seated with feet fully supported on a surface. During the recordings, the volunteers will be instructed to achieve relaxation to measure the resting state, and then they will be asked to perform an active movement of the affected lower limb.
Changes in cadence | Baseline and week 8 (after 24 sessions of intervention)
  An inertial sensor system (LegSys) will be placed above the malleolus in both lower limbs for assessing gait cadence. The patient will be asked to walk at their normal pace for a 10 (ten) metre length, if necessary with their assistive device.
Changes in stride length | Baseline and week 8 (after 24 sessions of intervention)
  An inertial sensor system (LegSys) will be placed above the malleolus in both lower limbs for assessing gait cadence. The patient will be asked to walk at their normal pace for a 10 (ten) metre length, if necessary with their assistive device.
Change in stride time | Baseline and week 8 (after 24 sessions of intervention)
  An inertial sensor system (LegSys) will be placed above the malleolus in both lower limbs for assessing gait cadence. The patient will be asked to walk at their normal pace for a 10 (ten) metre length, if necessary with their assistive device.
Change in swing phase | Baseline and week 8 (after 24 sessions of intervention)
  An inertial sensor system (LegSys) will be placed above the malleolus in both lower limbs for assessing gait cadence. The patient will be asked to walk at their normal pace for a 10 (ten) metre length, if necessary with their assistive device.
Change in stance phase | Baseline and week 8 (after 24 sessions of intervention)
  An inertial sensor system (LegSys) will be placed above the malleolus in both lower limbs for assessing gait cadence. The patient will be asked to walk at their normal pace for a 10 (ten) metre length, if necessary with their assistive device.
Change in double support | Baseline and week 8 (after 24 sessions of intervention)
  An inertial sensor system (LegSys) will be placed above the malleolus in both lower limbs for assessing gait cadence. The patient will be asked to walk at their normal pace for a 10 (ten) metre length, if necessary with their assistive device.
Change in stride velocity | Baseline and week 8 (after 24 sessions of intervention)
  An inertial sensor system (LegSys) will be placed above the malleolus in both lower limbs for assessing gait cadence. The patient will be asked to walk at their normal pace for a 10 (ten) metre length, if necessary with their assistive device.
Change in spasticity | Baseline, immediately after first session and week 8 (after 24 sessions of intervention)
  Modified Tardieu scale will be performed with volunteers in supine position, and the assessed lower limb extended on the stretcher. Passive stretching of the triceps surae will be applied with faster speed and then with slow speed from the position of maximum plantarflexion to the maximum possible dorsiflexion to determine the values of R1 (the angle of muscle reaction with fast speed stretch) and R2 (degrees of dorsiflexion reached with slow speed stretch).

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Intelangelo, MSc, Study Director — Universidad del Gran Rosario
Locations (1):
- Department of Physical Therapy, Neurofunctional Research Unit - UIN, University Center for Assistance, Teaching and Research - CUADI University of Gran Rosario, Rosario, Santa Fe Province, Argentina